CLINICAL TRIAL: NCT07375823
Title: Effects of Electrical Muscle Stimulation Applied Concurrently With Active Movement and Exercise Therapy in Cervical Radiculopathy: A Randomized Trial
Brief Title: Effects of Exercises and Electrical Current Application Aiming to Strengthen Neck and Shoulder Blades Muscles on Symptoms of a Pinched Nerve in the Neck
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European University of Lefke (Other)
Responsible Party: Principal Investigator, Zhanna Abdrakhmanova, Physiotherapist, European University of Lefke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAYEK057.12
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Cervical Radiculopathy; Cervical Radicular Pain; Neck Pain; Numbness; Paresthesia; Weakness, Muscle; Endurance
Keywords: cervical radiculopathy (CR); radicular pain; radicular symptoms; scapular dyskinesia; cervical deep flexors endurance (CDFE); cervical spine functional performance; electrical muscle stimulation; resistance training; superimposition
MeSH Terms: conditions — Radiculopathy; Neck Pain; Hypesthesia; Paresthesia; Muscle Weakness | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Voluntary Exercise (Active Comparator): Active therapeutic exercises prescription for neck and scapular region, including warm-up, strengthening and cool - down under supervision of a physiotherapist.
  Interventions: Procedure: Exercise Therapy
- Electrically Stimulated Exercise (Experimental): All of the therapeutic exercises prescription parameters for warm-up, strengthening and cool - down, including patient positioning, type of exercise, duration, frequency and intensity will be the same as in 'Voluntary Exercise'.
  For the intervention details, while 'Voluntary Exercise' will recieve only active exercises under supervision of the physiotherapist, in 'Electrically Stimulated Exercise' as a part of the strengthening protocol, electrical muscle stimulation unit will be applied over scapular region, bilaterally.
  Interventions: Procedure: Superimposition of electrical muscle stimulation on active movement

INTERVENTIONS:
Procedure: Exercise Therapy — Active therapeutic exercises prescription in face - to - face therapy sessions under supervision, for the duration of approximately 60 minutes per session.
  Therapy session will start with a warm - up including segmental stability exercise , i.e. deep cervical flexors training to improve neuromuscular coordination of the neck: Participant will do chin - tucks (cervical retraction and axial extension) for 2 sets of 5 seconds hold for 12 repetions, with between set rest interval of 2 minutes, in sitting.
  Next, participant will perform global stability exercises emphasizing flexor and extensor group musculature, with a gym ball, as a part of strengthening protocol.
  Lastly, as a cool -down, participant performs: pectoralis stretch, scalene stretch, suboccipitals stretch. Each position is held for 15 seconds and repeated 4 times for each muscle group bilaterally.
  Arms: Voluntary Exercise
Procedure: Superimposition of electrical muscle stimulation on active movement — EMS will be applied over scapular region, bilaterally. Electophysiological motor points of upper trapezius will be identified through surface mapping with a pen electrode to minimize limited spatial recruitment of motor units, that occurs due to poor electrodes placement.
  Reference electrode is placed at the antagonist muscle, i.e. insertion of lower trapezius over the medial end of spine of scapula. Self - adhesive, disposable electrodes (4pcs) will be allocated for each participant at the first session.
  Movements of the participants will be synchronized with the EMS impulses, i.e. motion intiation - ramp up, hold - on time, rest - off time. Since present systematic reviews contain low quality evidence and EMS parameters are highly heteregenous, choice of the parameters will be done activating slow - twitch endurance muscle fibers.
  Arms: Electrically Stimulated Exercise

SUMMARY:
Cervical Radiculopathy (CR) is an objective loss of sensory and/or motor function as a result of compression or irritation of the cervical spinal nerve root.

The individuals with CR present with findings indicating an altered neural control of the neck musculature, leaving the cervical spine vulnerable to reactive forces.

Thus, physical therapy options should mainly focus on improving muscle function of the neck.

Given the promising results of electrical muscle stimulation and exercise therapy in recent literature the proposed study is aimed to investigate the effects of exercise therapy with electrical muscle on cervical muscle function and see, if muscle control has any impact on CR findings.

A superiority, randomized trial, with 2 intervention groups and allocation ratio of 1:1. 50 students, at the age from 18 to 29, from healthcare - related departments of European University of Lefke, who are diagnosed with CR will be recruited in the study.

To assess neck muscle function - Deep Neck Flexors Endurance time (s) and Cervical Progressive Iso - inertial Lifting scores (kg) will be used. Pain (Numeric Rating Scale 0 -10) and Muscle strength (grades 0 -5) will be used to measure the impact on CR findings.

All of the therapeutic exercises prescription parameters for warm-up (deep cervical flexors training), strengthening (cervical and scapulo-thoracic resistance training) and cool - down (flexibility training), will be the same for both groups: 60 minutes per session, 2 days in a week, for 6 weeks. In total each participant will recieve 12 sessions.

For the intervention details, while 'Intervention Group 1' will recieve only active exercises under supervision of the physiotherapist, in 'Intervention Group 2' as a part of the strengthening protocol, EMS will be applied over scapular region, bilaterally.

DETAILED DESCRIPTION:
Cervical Radiculopathy (CR) is an objective loss of sensory and/or motor function as a result of conduction block in axons of a spinal nerve or its roots due to compression or irritation of the cervical spinal nerve root . Etiology is attributed to cervical foraminal compression in 70-75 % of cases due to anterior and posterior degenerative changes of the zygapophyseal joints, cervical spondylosis and reduction in disc height. The most common clinical manifestations of CR include sensory impairments (e.g. paresthesia), motor abnormalities (e.g. muscle weakness) and neck pain radiating to the arm.

It is a common diagnosis, incidence of which ranged between 0.832 - 1.79 per 1,000 person, and prevalence values ranged from 1.21 - 5.8 per 1,000 according to the latest epidemiological studies.

The incidence of neck pain was found to be high in college students: 48%-78%. What is more, the annual growth rate of cervical spondylosis in college students was twice that of the 50-year-old participants. A high incidence of neck pain among college students was associated with a heavy academic workload and the pressure of examinations, which may lead to the deformation of the neck and shoulders, as well as soft tissue damage.

In the meta-analysis of the college grade differences on neck pain in 2287 college students, it was shown that a higher probability and frequency of neck pain occurred at senior grade level. As can be seen from the review of existing literature, based on the incidence of neck pain, the potential of developing cervical radiculopathy is increasing at a younger age than was previously believed, with the peak age being 50 to 54 years. If left untreated, CR could lead to future disability and persistent functional impairments due to neural inflammation and edema, hypoxia and ischemia of structures.

However, despite the severity of the condition and the rapid incidence growth rate, there is still a lack of evidence in the area of conservative treatment, i.e. physiotherapy options. In previous studies, Electrical Muscle Stimulation (EMS) had no significant impact on pain relief, disability and patient satisfaction when used as an adjunct to cervical mobilization and manipulation, at post treatment, short-term and intermediate-term follow-up. Moreover, exercise treatment (ET) also consists of various interventions and is typically combined with drugs and other treatments, which make it difficult to determine the effects of a single intervention.

Nevertheless, results of more recent studies, are favoring application of EMS on various muscle groups, for example it was stated that EMS has significant effect on muscle strength of quadriceps and trunk extensors, similar results were also observed in the study assessing effects of EMS on upper extremity strength. Moreover, it was shown that neuromuscular electrical stimulation (NMES) induced a decrease of cortical activation during execution of hand movements, which indicates that application of NMES can increase the efficiency of the cerebral cortex during execution of motor tasks.

One should also consider that in the recent systematic review solitary ET directed on strengthening deep cervical flexors, scapulo - thoracic and upper extremity muscles had beneficial effect on pain and function at immediate post treatment and up to long-term follow-up. Moreover, strong evidence was found for effectiveness of deep cervical flexors (DCF) training on neuromuscular coordination of the neck, because it reduces the overactivation of the superficial muscles and improves the activation pattern of the cervical muscles.

It is also worth mentioning that, compared with the healthy adults, the individuals with CR have significantly smaller anterior displacements of the centers of mass and pressure, reduced muscle activity of the upper trapezius, sternocleidomastoid and splenius capitis muscles in response to all postural perturbations. Those findings are indicative of altered neural control of the neck musculature, leaving the cervical spine vulnerable to reactive forces.

Thus, physical therapy options for conservative management of CR should mainly focus on improving muscle function and neuromuscular control of the neck.

Given the promising results of EMS and ET, it is worth to investigate both in terms of neck muscle function. Thus, this research will try to do that.

Looking at the existing literature, training based on electrical muscle stimulation and voluntary muscle contraction has positive effects on muscle strength of various muscle groups, when applied in superimposition due to facilitation of additional muscle fibers recruitment.

However, superimposition of electrical stimulation on exercise was not assessed in the context of CR patients, who present with incomplete central activation levels and could favor from this kind of treatment, in terms of improving motor control. Additionally, restoring muscle balance in cervico - scapular region, adds to the proper neutral alignment of the cervical vertebrae, leading to increased intervertebral foraminal area, decreased nerve root compression and relieve of cervical radiculopathy symptoms.

Thus, the proposed study is aimed to investigate the effects of exercise therapy with electrical muscle stimulation and just exercise on cervical muscle function. Secondly, compare the effects of both therapy options. Lastly, see if improvement of neck muscle function would have and impact on cervical radiculopathy symptoms, in terms of pain and motor deficits.

ELIGIBILITY:
Inclusion Criteria:

* Student must be enrolled in the last 2 years of Bachelor degree or in Master's degree in one of the healthcare - related programs at the European University of Lefke;
* Age 18 - 29 years old;
* Neck pain of minimum 4 or more on numerical rating scale (0 - 10);
* Duration of symptoms 3 < months < 6, i.e. subacute symptoms with chronic/stable presentation;
* Has 1 or more of the following symptoms: paresthesia of 1 or both upper extremities at the level below elbow; pain radiating from neck to shoulder/arm/below elbow; feeling of weakness in 1 or both of the upper extremities, stiffness and/or tenderness and/or hyperalgesia in the cervical and/or upper thoracic area;
* Obtained "Cervical Radiculopathy" diagnosis from a physician, according to neurological examination findings: Positive cervical radiculopathy specific provocative tests (Spurling's Maneuver, Upper Limb Tension Test; Reduced Deep Tendon Reflexes of brachioradialis, biceps and triceps.

Exclusion Criteria:

* Any recent head/neck or shoulder trauma in the last 3 months;
* Received physiotherapy for neck - related complaints in the last 3 months;
* Received or currently receiving any kind of pharmacological intervention (muscle relaxants, NSAIDs, corticosteroids injections) in the last 3 months;
* Presents with symptoms favoring shoulder pathology: pain localized at the shoulder that worsens at night, positive Drop Arm Test, pain referral patterns are localized in the upper arm above elbow;
* Any recent surgeries to the neck, upper extremities within the last 6 months;
* Any diagnosed neurologic or musculoskeletal conditions that could mimic cervical radiculopathy, i.e. peripheral neuropathies of different origin, thoracic outlet syndrome medial/lateral epicondylitis, myofascial pain syndrome, etc.;
* Any cardiovascular (recent DVT, congestive heart failure), metabolic (diabetic polyneuropathy), neurologic (impaired consciousness, epilepsy), malignant conditions in which application of electrotherapy or exercises imposes risk on the patient;
* Presence of pregnancy;
* Active implants, e.g. cardiac pacemaker;
* Any skin lesions in the cervical and/or scapular region, i.e. infections, open - wounds;
* Refuses to participate in the study.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Deep Neck Flexors Endurance Test | From pre - treatment (at the enrollment stage) to post - treatment assessment after 6 weeks (12th session).
  To assess motor control of the neck, deep neck flexors endurance test will be used as a measure of neck muscle function. The reliability indexes suggest that the Deep Neck Flexors Endurance Test (DNFET )is an appropriate measure for group comparisons.
Cervical Progressive Iso - Inertial Lifting Evaluation | From pre - treatment (at the enrollment) to post - treatment assessment after 6 weeks (12th session).
  Cervical Progressive Iso - Inertial Lifting Evaluation is functional restoration measure in spinal disorders. The endurance test of the short neck flexors and the cervical PILE test can be regarded as appropriate instruments for measuring different aspects of neck muscle function in patients with non-specific neck pain. Moreover, the cervical PILE test - showed high inter-rater reliability and between-days repeatability out of 8 physical performance tests.

SECONDARY OUTCOMES:
Muscle Strength Assessment | From pre - treatment (at the enrollment) to post - treatment assessment at 6 weeks (after 12th session).
  Muscle strength testing of the Biceps Brachii and Deltoid had highest sensitivity, while Biceps Brachii and Triceps Brachii had highest specificity, with overall sensitivity being 61% compared to imaging and electromyographic studies in the diagnosis of Cervical Radiculopathy.
  Thus, muscle strength of biceps brachii, triceps brachii and deltoids will be used as an outcome measure in this study and assessed according to Manual Muscle Test grades 0 to 5.
  Muscle strength has been classified into 6 grades, from 0 being no evidence of muscle contraction, 1- palpatable muscle contraction and no range of motion, 2 - active movement throughout range of motion without gravity, 3 - active movement throughout range of motion against gravity and no other resistance, 4 - active range of motion against gravity and slight resistance, 5 - ability to maintain test position against gravity and maximal resistance.
Pain (Numeric Pain Rating Scale) | From pre - treatment (at enrollment stage) to post - treatment assessment at 6 weeks (after 12th session).
  The intensity of pain can be assessed by Numeric Rating Scale (NRS) in cases of Cervical Radiculopathy. The Numerical Rating Scale uses whole numbers from 0 to 10 along a line or a bar, with 0 indicating no pain and 10 being the most excruciating pain one has ever felt. 4 or 5 points (average pain intensity) on the 10 point scale are usually considered as an indication for physical therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Zhanna Abdrakhmanova, BSc in Physical Therapy, Principal Investigator — European University of Lefke; Nazemin Gilanlıoğulları, Asst. Prof. Dr., PhD in Rehabilitation, Study Chair — Faculty of Health Sciences, Vice Dean, European University of Lefke; Beraat Alptuğ, Asst. Prof. Dr., PhD in Physical Therapy, Study Chair — Head of the Department of Physiotherapy and Rehabilitation Faculty of Health Sciences European University of Lefke
Locations (1):
- European University of Lefke, Lefka, Cyprus

REFERENCES:
- [Background] Akesson I, Lundborg G, Horstmann V, Skerfving S. Neuropathy in female dental personnel exposed to high frequency vibrations. J Occup Environ Med. 1995;52(2): 116-23, http://dx.doi.org/10.1136/oem.52.2.116.
- [Background] Algarni AD, Al-Saran Y, Al-Moawi A, Bin Dous A, Al-Ahaideb A, Kachan athu SJ. The Prevalence of and Factors Associated with Neck, Shoulder, and Low-Back Pains among Medical Students at University Hospitals in Central Saudi Arabia. Pain Res Treat. 2017;2017:1235706. https://doi.org/ 10.1155/2017/1235706
- [Background] Alshami, A. M., & Bamhair, D. A. (2021). Effect of manual therapy with exercise in patients with chronic cervical radiculopathy: a randomized clinical trial. Trials, 22(1), 716. https://doi.org/10.1186/s13063-021-05690-y
- [Background] American College of Sports Medicine ACSM's for exercise testing and prescription, 10th edition, 2018
- [Background] Anekstein, Y., Blecher, R., Smorgick, Y., & Mirovsky, Y. (2012). What is the best way to apply the Spurling test for cervical radiculopathy?. Clinical orthopaedics and related research, 470(9), 2566-2572. https://doi.org/10.1007/s11999-012-2492-3
- [Background] Barsi, G.I., Popovic, D.B., Tarkka, I.M. et al. Cortical excitability changes following grasping exercise augmented with electrical stimulation. Exp Brain Res 191, 57-66 (2008). https://doi.org/10.1007/s00221-008-1495-5
- [Background] Boudreau, S.A., Falla, D. Chronic neck pain alters muscle activation patterns to sudden movements. Exp Brain Res 232, 2011-2020 (2014). https://doi.org/10.1007/s00221-014-3891-3
- [Background] Brage, K., Ris, I., Falla, D., Søgaard, K., & Juul-Kristensen, B. (2015). Pain education combined with neck- and aerobic training is more effective at relieving chronic neck pain than pain education alone - A preliminary randomized controlled trial. Manual Therapy, 20(5), 686-693. https://doi.org/10.1016/j.math.2015.06.003
- [Background] Carette S, Fehlings MG (2005) Clinical practice. Cervical radiculopathy. N Engl J Med 353(4):392-399
- [Background] Chan CWY. Neurophysiological basis underlying the use of resistance to facilitate movement. Physiother Can. 1984;36(6):335-341.
- [Background] Childress, M. A., & Becker, B. A. (2016). Nonoperative Management of Cervical Radiculopathy. American family physician, 93(9), 746-754.
- [Background] Coenen P, Kingma I, Boot CR, Twisk JW, Bongers PM, van Dieen JH. Cumulative low back load at work as a risk factor of low back pain: A prospective cohort study. J Oc cup Rehabil. 2013;23(1):11-8, http://dx.doi.org/10.1007/ s10926-012-9375-z.
- [Background] Cools AM, Declercq GA, Cambier DC, Mahieu NN, Witvrouw EE. Trapezius activity and intramuscular balance during isokinetic exercise in overhead athletes with impingement symptoms. Scand J Med Sci Sports. 2007; 17:25-33.
- [Background] Crawford RJ, Volken T, Schaffert R, Bucher T. Higher low back and neck pain in final year Swiss health professions' students: worrying susceptibilities identified in a multi-centre comparison to the national population. BMC Public Health. 2018;18(1):1188. https://doi.org/10.1186/ s12889-018-6105-2.
- [Background] Crochetiere WJ, Vodovnik L, Reswick JB: Electrical stimulation of skeletal muscle- a study of muscle as an actuator. Med Biol Eng 1967, 5:111-125
- [Background] de Koning, C. H., van den Heuvel, S. P., Staal, J. B., Smits-Engelsman, B. C., & Hendriks, E. J. (2008). Clinimetric evaluation of methods to measure muscle functioning in patients with non-specific neck pain: a systematic review. BMC musculoskeletal disorders, 9, 142. https://doi.org/10.1186/1471-2474-9-142
- [Background] Dirito, A. M., Abichandani, D., Jadhakhan, F., & Falla, D. (2024). The effects of exercise on neuromuscular function in people with chronic neck pain: A systematic review and meta-analysis. PloS one, 19(12), e0315817. https://doi.org/10.1371/journal.pone.0315817
- [Background] Doig, G. S., & Simpson, F. (2005). Randomization and allocation concealment: A practical guide for researchers. Journal of Critical Care, 20(2), 187-191. https://doi.org/10.1016/j.jcrc.2005.04.005
- [Background] Doucet BM, Lam A, Griffin L: Neuromuscular electrical stimulation for skeletal muscle function. Yale J Biol Med 2012, 85:201-215.
- [Background] Du, J., Zhang, L., Xu, C., & Qiao, J. (2021). Relationship Between the Exposure to Occupation-related Psychosocial and Physical Exertion and Upper Body Musculoskeletal Diseases in Hospital Nurses: A Systematic Review and Meta-analysis. Asian nursing research, 15(3), 163-173. https://doi.org/10.1016/j.anr.2021.03.003
- [Background] Falla, D., Jull, G., & Hodges, P. W. (2004). Feedforward activity of the cervical flexor muscles during voluntary arm movements is delayed in chronic neck pain. Experimental brain research, 157(1), 43-48. https://doi.org/10.1007/s00221-003-1814-9
- [Background] Gao, Y., Chen, Z., Chen, S., Wang, S., & Lin, J. (2023). Risk factors for neck pain in college students: A systematic review and meta-analysis. BMC Public Health, 23(1). https://doi.org/10.1186/s12889-023-16212-7
- [Background] Gellhorn E. Patterns of muscular activity in man. Arch Phys Med Rehabil. 1947;28:568-574.
- [Background] Gobbo, M., Maffiuletti, N. A., Orizio, C., & Minetto, M. A. (2014). Muscle Motor Point identification is essential for optimizing neuromuscular electrical stimulation use. Journal of NeuroEngineering and Rehabilitation, 11(1). https://doi.org/10.1186/1743-0003-11-17
- [Background] Gorce, P., & Jacquier-Bret, J. (2023). Global prevalence of musculoskeletal disorders among physiotherapists: A systematic review and meta-analysis. BMC Musculoskeletal Disorders, 24(1). https://doi.org/10.1186/s12891-023-06345-6
- [Background] Hagert, C.-G., Hagert, E., & Slutsky, D. (2008). Chapter 36: Manual Muscle Testing- A Clinical Examination Technique for Diagnosing Focal Neuropathies in the Upper Extremity. In Upper Extremity Nerve Repair: Tips and Techniques (pp. 451-457). essay, American Society for Surgery of the Hand. Retrieved from https://www.researchgate.net/publication/235979546
- [Background] Hanvold TN, Wærsted M, Mengshoel AM, Bjertness E, Twisk J, Veiersted KB. A longitudinal study on risk factors for neck and shoulder pain among young adults in the transition from technical school to working life. Scand J Work Environ Health. 2014;40(6):597-609. https://doi.org/10. 5271/sjweh.3437
- [Background] Harris KD, Heer DM, Roy TC, et al. Reliability of a measurement of neck flexor muscle endurance. Phys Ther 2005;85:1349-1355.
- [Background] Higgins, M., & Greer, C. (2025). Proprioceptive neuromuscular facilitation for the upper extremity and scapula: Review and update on rehabilitation of shoulder pathology. International Journal of Sports Physical Therapy, 20(9). https://doi.org/10.26603/001c.143176
- [Background] Honet JC, Puri K. Cervical radiculitis: treatment and results in 82 patients. Arch Phys Med Rehabil. 1976;57(1):12-16
- [Background] Hopewell S, Chan AW, Collins GS, Hróbjartsson A, Moher D, Schulz KF, et al. CONSORT 2025 Statement: updated guideline for reporting randomised trials. BMJ. 2025; 388:e081123. https://dx.doi.org/10.1136/bmj-2024-081123
- [Background] Horneij E, Holmström E, Hemborg B, Isberg PE, Ekdahl C. Inter-rater reliability and between-days repeatability of eight physical performance tests. AdvPhysiother. 2002;4:146-160.
- [Background] Iyer S, Kim HJ. Cervical radiculopathy. Curr Rev Musculoskelet Med. 2016;9(3):272-280. doi:10.1007/s12178-016-9349-4
- [Background] Jang, S. H., Jang, W. H., Chang, P. H., Lee, S. H., Jin, S. H., Kim, Y. G., & Yeo, S. S. (2014). Cortical activation change induced by neuromuscular electrical stimulation during hand movements: a functional NIRS study. Journal of neuroengineering and rehabilitation, 11, 29. https://doi.org/10.1186/1743-0003-11-29
- [Background] Jull, G. A., Falla, D., Vicenzino, B., & Hodges, P. W. (2009). The effect of therapeutic exercise on activation of the deep cervical flexor muscles in people with chronic neck pain. Manual Therapy, 14(6), 696-701. https://doi.org/10.1016/j.math.2009.05.004
- [Background] Kang M, Ragan BG, Park JH. Issues in outcomes research: an overview of randomization techniques for clinical trials. J Athl Train. 2008 Apr-Jun;43(2):215-21. doi: 10.4085/1062-6050-43.2.215. PMID 18345348
- [Background] Katsuura, Y., Bruce, J., Taylor, S., Gullota, L., & Kim, H. J. (2019). Overlapping, masquerading, and causative cervical spine and shoulder pathology: A systematic review. Global Spine Journal, 10(2), 195-208. https://doi.org/10.1177/2192568218822536
- [Background] Kemmler, W., Shojaa, M., Steele, J., Berger, J., Fröhlich, M., Schoene, D., von Stengel, S., Kleinöder, H., & Kohl, M. (2021). Efficacy of whole-body electromyostimulation (WB-Ems) on body composition and muscle strength in non-athletic adults. A systematic review and meta-analysis. Frontiers in Physiology, 12. https://doi.org/10.3389/fphys.2021.640657
- [Background] Kim DG, Chung SH, Jung HB. The effects of neural mobilization on cervical radiculopathy patients' pain, disability, ROM, and deep flexor endurance. J Back Musculoskelet Rehabil 2017;30:951-9.
- [Background] KISNER, C., COLBY, L. A., & BORSTAD, J. (2018). Therapeutic exercise: Foundations and techniques Carolyn Kisner, Lynn Allen Colby, John Borstad (7th ed.). F.A. Davis Company.
- [Background] Kleinrensink, G. J., Stoeckart, R., Mulder, P. G., Hoek, G., Broek, T., Vleeming, A., & Snijders, C. J. (2000). Upper limb tension tests as tools in the diagnosis of nerve and plexus lesions. Anatomical and biomechanical aspects. Clinical biomechanics (Bristol, Avon), 15(1), 9-14. https://doi.org/10.1016/s0268-0033(99)00042-x
- [Background] Koutedakis, Y., Frischknecht, R., Vrbová, G., Sharp, N. C., and Budgett, R. (1995). Maximal voluntary quadriceps strength patterns in Olympic overtrained athletes. Med. Sci. Sports Exerc. 27, 566-572. doi: 10.1249/00005768-199504000-00015
- [Background] Kroeling P, Gross A, Graham N, Burnie SJ, Szeto G, Goldsmith CH, Haines T, Forget M. Electrotherapy for neck pain. Cochrane Database of Systematic Reviews 2013, Issue 8. Art. No.: CD004251. DOI: 10.1002/14651858.CD004251.pub5
- [Background] Lee, M.-C., Ho, C.-S., Hsu, Y.-J., Wu, M.-F., & Huang, C.-C. (2023). Effect of 8-week frequency-specific electrical muscle stimulation combined with resistance exercise training on Muscle Mass, strength, and body composition in men and women: A feasibility and Safety Study. PeerJ, 11. https://doi.org/10.7717/peerj.16303
- [Background] Liang, L., Feng, M., Cui, X., Zhou, S., Yin, X., Wang, X., Yang, M., Liu, C., Xie, R., Zhu, L., Yu, J., & Wei, X. (2019). The effect of exercise on cervical radiculopathy. Medicine, 98(45). https://doi.org/10.1097/md.0000000000017733
- [Background] Lima LV, Abner TSS, Sluka KA. Does exercise increase or decrease pain? Central mechanisms underlying these two phenomena. J Physiol 2017;595:4141-50
- [Background] Lin, CC., Lin, CF., Hua, SH. et al. Chronic Neck Pain Affects Shoulder Muscle Activity and Postural Control During Functional Reach. J. Med. Biol. Eng. 41, 77-83 (2021). https://doi.org/10.1007/s40846-020-00591-y
- [Background] Lin, S. C., Lin, L. L., Liu, C. J., Fang, C. K., & Lin, M. H. (2020). Exploring the factors affecting musculoskeletal disorders risk among hospital nurses. PloS one, 15(4), e0231319. https://doi.org/10.1371/journal.pone.0231319
- [Background] Lindell O, Eriksson L, Strender LE. The reliability ofa 10-test package for patients with prolonged back and neck pain: could an examiner without formal medicaleducation be used without loss of quality? Amethodological study. BMC Musculoskelet Disord.2007;8:1-12
- [Background] Ludwig O, Berger J, Becker S, Kemmler W, Fröhlich M. 2019. The impact of whole-body electromyostimulation on body posture and trunk muscle strength in untrained persons. Frontiers in Physiology 10:1020 DOI 10.3389/fphys.2019.01020.
- [Background] Lundeberg, T., Lund, I., Dahlin, L., Borg, E., Gustafsson, C., Sandin, L., Rosén, A., Kowalski, J., & Eriksson, S. V. (2001). Reliability and responsiveness of three different pain assessments. Journal of rehabilitation medicine, 33(6), 279-283. https://doi.org/10.1080/165019701753236473
- [Background] Maicki T, Bilski J, Szczygieł E, Trąbka R. PNF and manual therapy treatment results of patients with cervical spine osteoarthritis. J Back Musculoskelet Rehabil. 2017;30(5):1095-1101. doi: 10.3233/ BMR-16971
- [Background] Mansfield, M., Smith, T., Spahr, N., & Thacker, M. (2020). Cervical spine radiculopathy epidemiology: A systematic review. Musculoskeletal Care, 18(4), 555-567. https://doi.org/10.1002/msc.1498
- [Background] Marco, B., Evans, D., Symonds, N., Peolsson, A., Coppieters, M. W., Jull, G., Löfgren, H., Zsigmond, P., & Falla, D. (2022). Determining the level of cervical radiculopathy: Agreement between visual inspection of pain drawings and magnetic resonance imaging. Pain Practice, 23(1), 32-40. https://doi.org/10.1111/papr.13147
- [Background] Martin-Gomez, C., Sestelo-Diaz, R., Carrillo-Sanjuan, V., Navarro-Santana, M. J., Bardon-Romero, J., & Plaza-Manzano, G. (2019). Motor control using cranio-cervical flexion exercises versus other treatments for non-specific chronic neck pain: A systematic review and meta-analysis. Musculoskeletal science & practice, 42, 52-59. https://doi.org/10.1016/j.msksp.2019.04.010
- [Background] Mayer TG, Barnes D, Kishino ND, Nichols G,Gatchel RJ, Mayer H et al. Progressive isoinertiallifting evaluation I. A standardized protocol andnormative database. Spine. 1988a;13:993-7.
- [Background] Muaidi Q, Shanb A. Prevalence causes and impact of work related musculoskeletal disorders among physical therapists. J Back Musculoskelet Rehabil. 2016;29(4):763-769. doi: 10.3233/BMR-160687.
- [Background] Olson LE, Millar AL, Dunker J, et al. Reliability of a clinical test for deep cervical flexor endurance. J Manip Physiol Ther 2006;29:134-138.
- [Background] Paillard T (2018) Training Based on Electrical Stimulation Superimposed Onto Voluntary Contraction Would be Relevant Only as Part of Submaximal Contractions in Healthy Participants. Front. Physiol. 9:1428. doi: 10.3389/fphys.2018.01428
- [Background] Panjabi MM, Cholewicki J, Nibu K, Grauer J, Babat LB, Dvorak J. Critical load of the human cervical spine: an in vitro experimental study. Clin Biomech (Bristol, Avon) 1998;13:11-17. doi: 10.1016/S0268-0033(97)00057-0
- [Background] Patel, P., Green, M., Tram, J., Wang, E., Murphy, M., Abd-Elsayed, A. a, & Chakravarthy, K. (2025). Latest advancements in transcutaneous electrical nerve stimulation (TENS) and electronic muscle stimulation (EMS): Revisiting an established therapy with new possibilities. Journal of Pain Research, Volume 18, 137-153. https://doi.org/10.2147/jpr.s493162
- [Background] Qin Y, Chen H, Liu X, Wu J, Zhang Y. 2022. Effects of whole-body electromyostimulation training on upper limb muscles strength and body composition in moderately trained males: a randomized controlled study. Frontiers in Public Health 10:982062 DOI 10.3389/fpubh.2022.982062.
- [Background] Rabiei M, Shakiba M, Dehgan-Shahreza HA, Talebzadeh M. Musculoskeletal disorders in dentists. International journal of occupational hygiene. 2012;4(1):36-40.
- [Background] Radhakrishnan K, Litchy WJ, O'Fallon WM, Kurland LT. Epidemiology of cervical radiculopathy. A population-based study from Rochester, Minnesota, 1976 through 1990. Brain. 1994;117(pt 2):325-335.
- [Background] Rafeemanesh, E., Omidi-Kashani, F., Chamani, A., & Allahdad, S. (2025). Occupational and Non-Occupational Risk Factors for Neck Pain in Dentists: A Systematic Review and Meta-Analysis. The archives of bone and joint surgery, 13(6), 307-322. https://doi.org/10.22038/ABJS.2024.78260.3604.
- [Background] Rafiq, S., Zafar, H., Gillani, S. A., Waqas, M. S., Liaqat, S., Zia, A., & Rafiq, Y. (2022b). Effects of Neurodynamic Mobilization on Health-Related Quality of Life and Cervical Deep Flexors Endurance in Patients of Cervical Radiculopathy: A Randomized Trial. BioMed research international, 2022, 9385459. https://doi.org/10.1155/2022/9385459
- [Background] Ren YC, Lin XG, Xie X, C YX. Status of cervical sub-health and its risk factors among college students. Chin J Sch Health. 2013;34(03):324-6+329. https://doi.org/10.16835/j.cnki.1000-9817.2013.03.023.
- [Background] Rubinstein, S. M., Pool, J. J., van Tulder, M. W., Riphagen, I. I., & de Vet, H. C. (2006). A systematic review of the diagnostic accuracy of provocative tests of the neck for diagnosing cervical radiculopathy. European Spine Journal, 16(3), 307-319. https://doi.org/10.1007/s00586-006-0225-6
- [Background] Schory, A., Bidinger, E., Wolf, J., & Murray, L. (2016). A SYSTEMATIC REVIEW OF THE EXERCISES THAT PRODUCE OPTIMAL MUSCLE RATIOS OF THE SCAPULAR STABILIZERS IN NORMAL SHOULDERS. International journal of sports physical therapy, 11(3), 321-336.
- [Background] Seddon HJ, Peripheral nerve injuries. In: The nerve injuries committee of the medical research council. London: Her Majesty's Stationery Office, 1954:1-451.
- [Background] Seyri KM, Maffiuletti NA. 2011. Effect of electromyostimulation training on muscle strength and sports performance. The Journal of Strength and Conditioning Research 33(1):70-75 DOI 10.1519/SSC.0b013e3182079f11.
- [Background] Szymanska J. Disorders of the musculoskeletal system among dentists from the aspect of ergonomics and prophylaxis. Ann Agric Environ Med. 2002;9(2):169-73.
- [Background] Tamburin, S., Paolucci, S., Magrinelli, F., Musicco, M., & Sandrini, G. (2016). The Italian Consensus Conference on pain in neurorehabilitation: Rationale and methodology. Journal of Pain Research, 311. https://doi.org/10.2147/jpr.s84646
- [Background] Thoomes, E. J., Scholten-Peeters, G. G., de Boer, A. J., Olsthoorn, R. A., Verkerk, K., Lin, C., & Verhagen, A. P. (2012). Lack of uniform diagnostic criteria for cervical radiculopathy in Conservative Intervention Studies: A systematic review. European Spine Journal, 21(8), 1459-1470. https://doi.org/10.1007/s00586-012-2297-9
- [Background] Viikari-Juntura E. Interexaminer reliability of observations in physical examinations of the neck. Phys Ther. 1987;67:1526-1532. doi: 10.1093/ptj/67.10.1526
- [Background] Walker, K. (1990). Chapter 72: Deep Tendon Reflexes. In Clinical Methods: The History, Physical, and Laboratory Examinations. (3rd ed.). essay.
- [Background] WHO guidelines on physical activity and sedentary behaviour. (2020). World Health Organization.
- [Background] Wong, J. J., Côté, P., Quesnele, J. J., Stern, P. J., & Mior, S. A. (2014). The course and prognostic factors of symptomatic cervical disc herniation with radiculopathy: A systematic review of the literature. The Spine Journal, 14(8), 1781-1789. https://doi.org/10.1016/j.spinee.2014.02.032
- [Background] Woods BI, Hilibrand AS. Cervical radiculopathy: epidemiology, etiology, diagnosis, and treatment. J Spinal Disord Tech. 2015;28(5):E251-9. https://doi.org/10.1097/BSD.0000000000000284
- [Background] YEŞİLYURT, M., & FAYDALI, S. (2020). Ağri Değerlendi̇rmesi̇nde Tek Boyutlu ölçekleri̇n Kullanimi. Journal of Anatolia Nursing and Health Sciences. https://doi.org/10.17049/ataunihem.508877
- [Background] Yousif, M. S., Occhipinti, G., Bianchini, F., Feller, D., Schmid, A. B., & Mourad, F. (2025). Neurological examination for cervical radiculopathy: A scoping review. BMC Musculoskeletal Disorders, 26(1). https://doi.org/10.1186/s12891-025-08560-9
- [Background] Zhao Jie Wu, Kunwei HW, Xiaoyu Hu, Xianyue Z. Influencing factors and preventive measures of spondylosis in college students. Healthmust Readmagazine. 2020;22:244.